CLINICAL TRIAL: NCT06072911
Title: Continence, Sexual and Metabolic Health Programming to Promote Prostate Cancer Wellness for Life (CONTROL4LIFE)
Brief Title: Continence, Sexual Function, Fitness and the Health of Men After Surgery for Prostate Cancer
Acronym: CONTROL4LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREBA.CC-23-0207
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Incontinence; Metabolic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Zelen design with randomization
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be randomized after the baseline assessment and will have the option to take part in an additional exercise intervention component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pelvic floor exercise program and general exercise programming
  Interventions: Behavioral: Pelvic floor exercise program; Behavioral: General exercise
- Control (Active Comparator): Pelvic floor exercises and standard care (physical activity counseling)
  Interventions: Behavioral: Pelvic floor exercise program; Behavioral: Physical Activity Counseling

INTERVENTIONS:
Behavioral: Pelvic floor exercise program — General exercises will be prescribed along with a specialized pelvic floor program
Behavioral: General exercise — A general progressive resistance exercise program
  Arms: Intervention
Behavioral: Physical Activity Counseling — Advice on increasing physical activity
  Arms: Control

SUMMARY:
The Continence, Sexual and Metabolic Health (CONTROL 4 LIFE) study will evaluate the recovery of continence, sexual function, and health outcomes in individuals who have undergone surgery for prostate cancer. The purpose of this study is to better understand the timelines of recovery for these outcomes after surgery for prostate cancer. As part of this study, all participants will receive resources offered by Alberta Health Services regarding pre- and post-prostatectomy care, including information on pelvic floor exercises. Through the CONTROL 4 LIFE study, the investigators will also be evaluating outcomes related to physical activity, fitness and quality of life. These assessments will enable the investigators to better understand how well and how long it takes for individuals to recover after surgery for prostate cancer.

DETAILED DESCRIPTION:
The investigators aim to conduct a trial examining the feasibility and the effects of a combined pelvic health rehabilitation and exercise program that can be delivered both in-person and virtually in individuals who have been treated with prostatectomy for prostate cancer. This hybrid format will support equitable program delivery regardless of location of residence. To address issues faced by men with prostate cancer, the investigators propose an intervention (offered virtually and in-person) that includes: 1) online education to support continence, sexual and overall health; 2) a group exercise fitness program that considers the needs and restrictions specific to the early post-prostatectomy surgical period, and 3) functional and intensive pelvic floor muscle exercise retraining to promote continence and sexual recovery.

Main objectives of this study

1. Determine the feasibility, defined as the acceptability and appropriateness, of a combined pelvic health rehabilitation and exercise fitness program that can be delivered both in-person and virtually.
2. Determine the effects of the program on the primary outcome measure of urinary continence in comparison with usual care.

Secondary objectives of this study

1. To determine the effects of the program on cardiometabolic indicators in comparison with usual care.
2. To determine the effects of the program on general fitness, secondary outcomes of urinary continence, sexual function, self-efficacy, and cancer symptom burden, in comparison with usual care.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of prostate cancer (stage I to IV);
* be scheduled for a prostatectomy surgery (any surgical approach);
* have no restriction to participate in at least mild levels of physical activity, as confirmed by the Physical Activity Readiness Questionnaire (PAR-Q+);
* speak and understand English.
* adult: 18 years of age or older
* optional exercise component: willing and able to commit to the 12-week intervention

Exclusion Criteria:

* have any medical conditions that may interfere with continence (i.e. neurological diseases);
* have any contraindications to exercise testing or training;
* have recent (>6 months) modifications to any medication aiming to reduce urinary incontinence (i.e. Myrbetric);
* do not have regular access to the internet and a smart device or a computer at home/ at their community center;
* are already receiving a pelvic floor exercise program through a pelvic floor physical therapist from their community.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Completion Rate | Final assessment at one year
  The number of participants completing the study including all planned outcomes

SECONDARY OUTCOMES:
Recruitment rate | One year
  Percentage of participants who are eligible and agree to participate
Adherence rate | Post-intervention: 12 weeks
  Adherence to the intervention components
24-hour pad test | 24 hours at two time points: immediate post surgery and 12 weeks
  Mean: Individual's urine loss by measuring weight (grams) of an absorbent pad
Expanded Prostate Cancer Index Composite for Clinical Practice | One-year
  16-questions: urinary function, sexual and erectile function, bowel and hormonal function; Scores: 0 (no symptoms) to 60 (most severe symptoms); Higher scores indicate worse functioning
International Consultation on Incontinence Questionnaire | One-year
  13 questions: occurrence and bother of lower urinary tract symptoms, quality of life; Range of scores: 0-20 voiding subscale; 0-20 incontinence symptoms; Higher scores indicate worse functioning
36-Item Short Form Survey | One-year
  Quality of life measure: Items are scored 0-100 (percentage of total possible score): Higher scores equal better quality of life
Edmonton Symptom Assessment Scale | One year
  11-item ordinal scale; Range 0-60; with higher scores indicating higher symptom burden
Self-efficacy Questionnaire: Incontinence | One year
  6 item ordinal scale: Range 0-60; Higher scores indicating higher self-efficacy
Grip Strength | 12 weeks
  Dyanometer: mean in kgs
Lower body strength | 12-weeks
  Sit-to-stand: mean number completed in 30 seconds
Upper limb mobility | 12 weeks
  Shoulder Range of Motion: mean value in degrees
Flexibility | 12-weeks
  Sit and reach: mean value in cm
Balance | 12-weeks
  One-leg stance test: mean time in seconds
Walking endurance | 12-weeks
  Six-minute walk test: mean distance in metres
Body Mass Index | 12-weeks
  Height and weight will be combined to calculate BMI: mean: weight in kilograms divided by height in metres squared
Glucose | 12-weeks
  mmol/L (mean value)
Insulin level | 12-weeks
  mmol/L (mean value)
Lipid profile | 12-weeks
  Cholesterol level: mg/dL (mean value)
Hemoglobin A1c | 12-weeks
  Value in percentage (mean value)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Hoy, MD, Principal Investigator — University of Alberta; Howard Evans, MD, Principal Investigator — University of Alberta; Margaret McNeely, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be housed on the University of Alberta's Dataverse
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following completion of the study and primary publication.

REFERENCES:
- [Derived] Bernard S, Evans H, Hoy NY, Suderman K, Cameron B, Sexsmith J, Kinnaird A, Rourke K, Dean L, Pituskin E, Usmani N, Tandon P, McNeely ML. Control4Life: A randomized controlled trial protocol examining the feasibility and efficacy of a combined pelvic health rehabilitation and exercise fitness program for individuals undergoing prostatectomy. Contemp Clin Trials. 2024 Apr;139:107482. doi: 10.1016/j.cct.2024.107482. Epub 2024 Feb 29. PMID 38431130